CLINICAL TRIAL: NCT01989767
Title: Application of Psychiatric Knowledge in the Rehabilitation Process in Return to Work.
Acronym: PKRW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hans Joergen Soegaard (Other)
Responsible Party: Sponsor-Investigator, Hans Joergen Soegaard, M.D., consultant, prof., ph.d., Region MidtJylland Denmark
Organization: Region MidtJylland Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sickness absence 2
Record Dates: First submitted 2013-11-10; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Mental Disorders
Keywords: sickness absence; rehabilitation; mental disorders; screening
MeSH Terms: conditions — Mental Disorders | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator): Rehabilitation as usual
  Interventions: Behavioral: control Rehabilitation as usual
- education (Experimental): education of rehabilitation officers in psychiatric topics plus rehabilitation as usual
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: control Rehabilitation as usual — Rehabilitation as usual
  Arms: control
Behavioral: education — Education as add on to to rehabilitation as usual
  Arms: education

SUMMARY:
The hypothesis was that education of rehabilitation officers who were responsible for rehabilitation back to work for sick-listed individuals in screening for mental disorders and psychiatric topics would increase the rate of return to work and reduce the number of sicklisted days

ELIGIBILITY:
Inclusion Criteria:

* sick-listed and belonging to the case-load of rehabilitation officers who participated in the intervention

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
rate of return to work | 1 year
  The rate of return to work was estimated by Poisson regression and Cox regression based on the duration from the date being sicklisted until the date of return to normal work.

SECONDARY OUTCOMES:
number of sickness absence days | ½ year
  After eight weeks of continuous sickness absence the number of sickness absence days within ½ year was counted

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Research Unit West, Regional Psychiatric Services West, Herning, Denmark